CLINICAL TRIAL: NCT04408183
Title: Efficacy, Safety, and Tolerability of GLS-1200 Topical Nasal Spray in the Prevention of Incident Confirmed, Symptomatic SARS-CoV-2 Infection
Brief Title: GLS-1200 Topical Nasal Spray to Prevent SARS-CoV-2 Infection (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer enrolling
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: T2R-002
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: SARS-CoV 2; Infection
Keywords: COVID-19
MeSH Terms: conditions — Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLS-1200 (Experimental): 1 mL of GLS-1200 per nostril, TID
  Interventions: Drug: GLS-1200
- 0.9 %Saline (Placebo Comparator): 1 mL of 0.9% Saline per nostril, TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLS-1200 — GLS-1200 is given as a nasal spray using an atomizer
  Arms: GLS-1200
Drug: Placebo — Placebo is given as a nasal spray using an atomizer
  Arms: 0.9 %Saline

SUMMARY:
This clinical trial will evaluate the safety, tolerability and effectiveness of topical GLS-1200 nasal spray to reduce the incidence of confirmed, symptomatic SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This Phase II randomized, placebo-controlled, double-blind study will assess whether topical GLS-1200 applied via nasal spray atomizer is well-tolerated and can reduce the incidence of confirmed SARS-CoV-2 infection. Subjects will be randomized to either the GLS-1200 or placebo group in a 2:1 ratio with a target enrollment of 225 subjects. Subjects will self-administer study drug three times daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide informed consent
* Able and willing to comply with study procedures
* Able and willing to utilize an approved form of pregnancy prevention for women of child bearing potential through to the end of treatment

Exclusion Criteria:

* Know allergy to quinine, quinidine, or mefloquine
* Confirmed prior positive test for SARS-CoV-2
* Treatment within the past 2 weeks with chloroquine, hydroxychloroquine, or remdesivir
* Pregnancy or documentation of pregnancy by pre-treatment urine test or breast feeding or plans to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sinus and Nasal Specialists of Louisiana, Baton Rouge, Louisiana
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Conroe Willis Medical Reasearch, Conroe, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLS-1200 | 0.9 %Saline
Started | 123 | 61
Completed | 112 | 59
Not Completed | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLS-1200 | 0.9 %Saline | Total
Number analyzed (Participants) | 123 | 61 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 58 | 167
  >=65 years | 14 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.81) | 41.3 (12.99) | 43.9 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 40 | 121
  Male | 42 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 118 | 58 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 79 | 33 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 38 | 19 | 57
Region of Enrollment [Number; unit: participants]
  United States | 123 | 61 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number Serious Adverse Events as Assessed by CTCAE v5.0
Time Frame: Through 4 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GLS-1200 | 0.9 %Saline
Number analyzed (Participants) | 123 | 61
Participants | 0 | 0

2. Primary Outcome: Incidence of SARS-CoV-2 Infection, Confirmed by PCR Relative to Treatment Group
Time Frame: Through 4 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GLS-1200 | 0.9 %Saline
Number analyzed (Participants) | 123 | 61
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through 4 weeks of treatment.
Arm/Group | GLS-1200 | 0.9 %Saline
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/61
Other Adverse Events (participants affected / at risk) | 41/123 | 21/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLS-1200 (N=123) | 0.9 %Saline (N=61)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Headache (Nervous system disorders) | 10 (10) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04408183/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04408183/SAP_001.pdf